CLINICAL TRIAL: NCT06137417
Title: Role of PET/CT in Peritoneal Deposits Assessment
Status: Not yet recruiting | Type: Observational
Sponsor: Aya Khaled Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Aya Khaled Mahmoud, assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: PET CT peritoneal deposits
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Peritoneal Metastases
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PET/CT — • Suspected patients known to have a primary malignant tumour, patients with metastasis of unknown primary and had incidental peritoneal lesions.

SUMMARY:
• Suspected patients known to have a primary malignant tumour, patients with metastasis of unknown primary and had incidental peritoneal lesions and will do PET/CT for assessment of peritoneal deposits

DETAILED DESCRIPTION:
Suspected patients known to have a primary malignant tumour, patients with metastasis of unknown primary and had incidental peritoneal lesions and will do PET/CT for assessment of peritoneal deposits. we will find its diagnostic role.

ELIGIBILITY:
Inclusion Criteria:

* • Suspected patients known to have a primary malignant tumour, patients with metastasis of unknown primary and had incidental peritoneal lesions.

Exclusion Criteria:

* • Patients unable to sit calm without movement during imaging.

  * Severely ill patients.
  * Patients unable to sleep in a fixed position for 20 minutes.
  * Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Suspected patients known to have a primary malignant tumour, patients with metastasis of unknown primary and had incidental peritoneal lesions and will do PET/CT for assessment of peritoneal deposits
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
role of pet/ct in peritoneal deposits assessment | 2 years
  Suspected patients known to have a primary malignant tumour, patients with metastasis of unknown primary and had incidental peritoneal lesions and will do PET/CT for assessment of peritoneal deposits

REFERENCES:
- [Background] Dawson H, Kirsch R, Messenger D, Driman D. A Review of Current Challenges in Colorectal Cancer Reporting. Arch Pathol Lab Med. 2019 Jul;143(7):869-882. doi: 10.5858/arpa.2017-0475-RA. Epub 2019 Jan 23. PMID 30672337
- [Background] Husain A, Chi DS, Prasad M, Abu-Rustum N, Barakat RR, Brown CL, Poynor EA, Hoskins WJ, Curtin JP. The role of laparoscopy in second-look evaluations for ovarian cancer. Gynecol Oncol. 2001 Jan;80(1):44-7. doi: 10.1006/gyno.2000.6036. PMID 11136568
- [Result] Patel CM, Sahdev A, Reznek RH. CT, MRI and PET imaging in peritoneal malignancy. Cancer Imaging. 2011 Aug 24;11(1):123-39. doi: 10.1102/1470-7330.2011.0016. PMID 21865109